CLINICAL TRIAL: NCT02919748
Title: Choral Singing For the Prevention of Dementia: A Randomized Controlled Trial
Brief Title: Choral Singing For the Prevention of Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Agency for Science, Technology and Research (Other); Nanyang Technological University (Other); University of Cambridge (Other); Ministry of Health, Singapore (Other Government)
Responsible Party: Principal Investigator, Feng Lei, Dr, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NUS-IRB: B-14-304
Record Dates: First submitted 2016-09-19; First posted 2016-09-29 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Dementia; Cognitive Decline
Keywords: dementia; cognitive decline; choral singing; health education program; randomized controlled trial
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention arm (Experimental): Choral Singing
  Interventions: Other: Choral Singing
- Control arm (Active Comparator): General Health Education Program and Group Activities
  Interventions: Other: Health Education Program

INTERVENTIONS:
Other: Choral Singing — Weekly sessions at 1 hour of choral singing.
  Arms: Intervention arm
Other: Health Education Program — Weekly session at 1 hour of health education talk and group activities
  Arms: Control arm

SUMMARY:
To evaluate the efficacy of choral singing in the prevention of dementia and examine the underlying mechanisms using Magnetic Resonance Imaging (MRI) technique and a panel of peripheral biomarkers in venous blood and urine. The investigators hypothesize that Choral singing could prevent cognitive decline among community-dwelling elderly who are at high risk of dementia. The underlying neural mechanisms involve the changes in brain structure and function that can be quantified using MRI technique. The changes in cognitive outcomes will be accompanied by observable changes from a panel of carefully selected peripheral biomarkers.

DETAILED DESCRIPTION:
Cognitive function declines with advancing age and the prevalence and incidence of dementia rises dramatically in later life. Impaired cognitive function limits one's ability to work, live and socialize, and represent a major obstacle for active aging. Data from Asian countries showed a clear role of cognitive function in contributing to functional disability independent of physical health. How to maintain good cognitive health in the later stage of life is an important and challenging question that requires well-founded research with good applicability. With no cure for dementia in sight presently, it is vitally important to find effective preventive measures. Candidates and potential avenues for intervention should be carefully evaluated in well-designed randomized controlled trials (RCT). Here the investigators propose choral singing as a novel approach for the prevention of cognitive decline and dementia; the investigators plan to test the hypothesized efficacy in a RCT based on a selected group of senior Singaporeans from the Jurong Area. This proposed research is built on a growing body of research evidence on the role of choral singing in health promotion and psychological wellbeing; and the fact that no trial has tested the potential effectiveness of choral singing in delaying cognitive decline and the onset of dementia.

The plasticity of the brain forms the scientific basis for the potential efficacy of choral singing in preventing cognitive decline and the incidence of dementia. It is well known that participating in various cognitive, social and productive activities is associated with improved cognitive function and lower risk of dementia. The protective effects on cognition may be particularly effective for certain subgroups. For example, analysis of local data showed that among the single and widowed elderly, an increase in social engagement was associated with a lower risk of cognitive impairment: compared with subjects in the lowest tertile of social engagement scores, the adjusted Odds Ratio (OR) of cognitive impairment was 0.50 for subjects in the second or the third tertile.

Data from previous clinical trials support that cognitive training is effective in improving cognitive function or delaying cognitive decline in the elderly. Functional gains from cognitive training have been reported to last up to five years, with a meta-analysis demonstrating that the protective effects of cognitive training on cognition in healthy elderly can persist years after training. In Singapore, a brain-computer interface based cognitive training system showed promise in improving memory and attention in healthy elderly. Specifically, the training led to significant improvement in immediate memory (p = 0.038), visuospatial/constructional (p = 0.014), attention (p = 0.039), and delayed memory (p<0.001) scores. However, cognitive training based on human trainer or brain-computer interface are expensive and hence the applicability as a preventive in real world setting for the general population is largely limited. Participants of such trainings also may not be able to maintain lasting interest and motivation. Given those considerations, relatively cost-effective and captivating methods are urgently needed and we believe choral singing is a promising candidate.

In Singapore, there are more than 200 school choirs. Most universities and tertiary education institutions have choirs developed as an expressive art form. Furthermore, there are numerous church choirs who sing with spiritual passion, and the professional choruses who are selected to sing and to perform. The existing resource can be tapped on in the future for large scale interventional initiative once solid data of its efficacy are produced from rigorously designed clinical studies.

In this collaborative research project that involves experts from multiple disciplines, the investigators propose to conduct a randomized clinical trial to examine the clinical efficacy of choral singing in the prevention of cognitive decline and dementia. As a cognitive stimulating activity, choral singing involves cognitive processes such as attention, memory, executive function and language. As a social activity, choral singing consists of group interactions which cultivate the feeling of being part of a meaningful community. Prior studies have demonstrated that situations and activities involving synchrony with others induces feelings of closeness and affiliation, and bolsters coordination with synchronization partners. Increased prosociality and conformity produced by synchrony may also be applied to other people more generally, even those who were not synchronization partners. Moreover, synchrony and affiliative orientations also share a bi-directional relationship, such that individuals who are more prone to prosocial tendencies are more likely to synchronize with others. As a physical exercise, choral singing requires the involvement of more than 100 muscles; it helps to improve lung function and circulation, promotes superior posture, and boost balance and resistance. Choral singing also requires the choristers to cooperate with each other, the discipline of listening to blend with fellow singers and need persistently hard work to stay on par with the level of other singers. All the above may contribute to long term cognitive benefits of choral singing.

Although theoretically plausible, the effectiveness of choral singing in preventing cognitive decline and dementia has not been studied scientifically. This proposed study will fill an important knowledge gap. The investigators aim to produce firm data on two year efficacy of choral singing in preventing cognitive decline and this will form the evidence base for further research and future interventional initiative.

ELIGIBILITY:
Inclusion Criteria:

1. Community-living elderly aged 60 years and above, and
2. Subjective cognitive complaints based on self-report, or
3. Objective cognitive impairment based on neuropsychological test scores (Z score < 0 and >-1.5), or
4. Multiple risk factors of dementia such as family history, depression, etc., and
5. Not demented: Clinical Dementia Rating (CDR) global score=0

Exclusion Criteria:

1. Any terminal illness, OR
2. Stroke, OR
3. Aphasia, OR
4. Marked hearing impairment, OR
5. Participating in another interventional study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes in cognitive performance | Baseline, 1 year, 2 year
  Measured using a composite cognitive test score based on results from a battery of 6 cognitive tests that measures the performance on multiple cognitive domains. The composite cognitive test score (CCTS) will be calculated as the average of Z scores standardised to the baseline mean and standard deviation of trial participants, with higher scores representing better cognitive performance.

SECONDARY OUTCOMES:
Changes in brain structure and function | Baseline, 1 year, 2 year
  Measured using brain magnetic resonance imaging (MRI)
Changes in biological markers | Baseline, 1 year, 2 year
  Measured using biological sampling
Depressive symptoms | Baseline, 6 month, 1 year, 2 year
  Measured using the Geriatric Depression Scale (GDS-15)
Anxiety symptoms | Baseline, 6 month, 1 year, 2 year
  Measured using the Geriatric Anxiety Inventory (GAI)
Stress | Baseline, 6 month, 1 year, 2 year
  Measured using the Perceived Stress Scale (PSS)
Sleep quality | Baseline, 6 month, 1 year, 2 year
  Measured using the Pittsburgh Sleep Quality Index (PSQI)
Neuropsychiatric symptoms | Baseline, 6 month, 1 year, 2 year.
  Measured using the Neuropsychiatric Inventory (NPI)
Changes in Rey Auditory Verbal Learning Test | Baseline, 1 year, 2 year
  Measured using Rey Auditory Verbal Learning Test (RAVLT)
Changes in Digit Span | Baseline, 1 year, 2 year
  Measured using Digit Span Task
Changes in Block Design | Baseline, 1 year, 2 year
  Measured using Block Design Test
Changes in Color Trails | Baseline, 1 year, 2 year
  Measured using Color Trails tests
Changes in Symbol Digit Modality | Baseline, 1 year, 2 year
  Measured using Symbol Digit Modality Test (SDMT)
Changes in Boston Naming | Baseline, 1 year, 2 year
  Measured using Boston Naming Test
Severity of symptoms of dementia | Baseline, 1 year, 2 year
  Measured using the Clinical Dementia Rating (CDR)
Changes in Mini-Mental State Examination | Baseline, 6 month, 1 year, 2 year
  Measured using the Mini-Mental State Examination (MMSE)
Changes in Montreal Cognitive Assessment | Baseline, 6 month, 1 year, 2 year
  Measured using the Montreal Cognitive Assessment (MoCA)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Feng, Medicine, Principal Investigator — National University of Singapore
Locations (1):
- TaRA@JP, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feng L, Ng TP, He Y, Li C, Kua EH, Zhang M. Physical Health and Cognitive Function Independently Contributed to Functional Disability among Chinese Older Adults: Data from Two Asian Metropolises. J Aging Res. 2011;2011:960848. doi: 10.4061/2011/960848. Epub 2011 Sep 14. PMID 21941656
- [Background] Feng L, Ng XT, Yap P, Li J, Lee TS, Hakansson K, Kua EH, Ng TP. Marital Status and Cognitive Impairment among Community-Dwelling Chinese Older Adults: The Role of Gender and Social Engagement. Dement Geriatr Cogn Dis Extra. 2014 Oct 14;4(3):375-84. doi: 10.1159/000358584. eCollection 2014 Sep. PMID 25473404
- [Background] Wu DX, Feng L, Yao SQ, Tian XF, Mahendran R, Kua EH. The early dementia prevention programme in Singapore. Lancet Psychiatry. 2014 Jun;1(1):9-11. doi: 10.1016/S2215-0366(14)70233-0. Epub 2014 Jun 4. No abstract available. PMID 26360390
- [Derived] Ng TKS, Lim ZH, Todd M, Sun F, Ray K, Qi X, Guo J, Ye KX, Maier AB, Mahendran R, Lee Gan G, Tsakok M, Kua EH, Feng L. Effects of choral singing on depression and anxiety in older adults: A randomized controlled trial. J Psychiatr Res. 2025 Aug;188:162-168. doi: 10.1016/j.jpsychires.2025.05.061. Epub 2025 May 26. PMID 40449223
- [Derived] Tan J, Tsakok FHM, Ow EK, Lanskey B, Lim KSD, Goh LG, Tan CH, Cheah IK, Larbi A, Foo R, Loh M, Wong CKY, Suckling J, Li J, Mahendran R, Kua EH, Feng L. Study Protocol for a Randomized Controlled Trial of Choral Singing Intervention to Prevent Cognitive Decline in At-Risk Older Adults Living in the Community. Front Aging Neurosci. 2018 Jul 10;10:195. doi: 10.3389/fnagi.2018.00195. eCollection 2018. PMID 30042673